CLINICAL TRIAL: NCT04463589
Title: Factors Associated With the Evolution of Presenteeism Under Biotherapy in Severe Asthma
Brief Title: Presenteeism in Severe Asthma Treated by Biotherapyasthma
Acronym: PRESATHMA
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_36; 2020-A00085-34 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-07-02; First posted 2020-07-09 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2023-12

CONDITIONS: Asthma
Keywords: Severe Asthma; Presenteism; Asthma burden; Biotherapy; Quality of life
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe asthma is a condition characterized by a lower sensitivity to high doses of inhaled corticosteroids combined with a second controller, most often a long-acting bronchodilator. It concerns approximately 5% of asthmatics. Treatment failure and co-morbidities induced by systemic corticosteroid therapy can cause debilitating dyspnea, limited physical activity, and impaired quality of life. Severe asthma could therefore be associated with major presenteeism, defined as the presence of an employee at work despite his health issues and which implies a limitation of the employee's productive capacity. Uncontrolled asthma and co-morbidities of asthma have been shown to be associated with a decrease in work productivity that includes absenteeism and presenteeism. Although there is little data, a recent study found a decline in work productivity in severe asthma. Various factors associated with presenteeism could be involved, such as asthma control, frequency and severity of exacerbations, comorbidities, or treatments.

Biotherapies targeting the signaling pathways involved in airway inflammation improve asthma control, decrease the frequency of asthma exacerbations which are major determinants of quality of life, improve lung function, and allow oral steroid sparing. Biotherapies could therefore be associated with a decrease in presenteeism.

The objective of the study is to describe the evolution of presenteeism at work, evaluated by the WPAI: Asthma, after 6 months of treatment by biotherapy and to identify factors associated with this evolution

ELIGIBILITY:
Inclusion Criteria:

* Severe asthma defined as the use of a high doses of inhaled corticosteroids combined with a second controller (GINA 4) and / or oral corticosteroid therapy > 50% of the year
* Eligible for biotherapy according to the investigator's decision
* Holders of an employment contract for at least 8 days
* Written non-opposition to participate in the study after information
* Social protection affiliation

Exclusion Criteria:

* Existence of another chronic pulmonary disease (bronchiectasis, COPD, diffuse interstitial lung disease, neuromuscular pathology, etc.) or cardiac (cardiac rhythm disorder, ischemic heart disease, etc.) significant according to the investigator's judgment
* Psychiatric disorder
* Pregnancy
* Persons under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe asthmatic patients starting a biotherapy
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Change in presenteeism | At 6 months
  Change Questionnaire Work Productivity and activity impairment : Asthma (WPAI : Asthma) - question 5 (Q5) after 6 months of biotherapy The WPAI-question 5 ranges from 0 to 10, a higher score meaning a worse outcome

SECONDARY OUTCOMES:
Correlation between the WPAI : Asthma- Q5 score and the ACQ-6 score | at baseline
  Association between presenteeism and asthma control Asthma Control Questionnaire (ACQ) is simple questionnaire to measure the adequacy of asthma control and change in asthma control, 7-point scale (0=no impairment, 6= maximum impairment for symptoms and rescue use; and 7 categories for FEV1%)
Correlation between the WPAI : Asthma- Q5 score and the mMRC score | at baseline
  Association between presenteeism and exercise dyspnea at baseline the mMRC (Modified Medical Research Council) Dyspnea Scale,The 1-5 stage scale is used alongside the questionnaire to establish clinical grades of breathlessness.
Correlation between the WPAI : Asthma- Q5 score and FEV1, la FVC and RV. | at baseline
  Association between presenteeism and airways obstruction at baseline
Correlation between the WPAI : Asthma- Q5 score and the STAI-Y2 score | at baseline
  Association between presenteeism and anxiety at baseline tate-Trait Anxiety Inventory, STAI-Y2 (STAI-Y2), consists of 20 sentences assessing the subject's usual emotional state.Each answer to an item in the STAI-Y is scored from 1 to 4, with 1 indicating the lowest degree of anxiety and 4 the highest degree of anxiety.
Correlation between the WPAI : Asthma- Q5 score and the Nijmegen score | at baseline
  Association between presenteeism and hyperventilation symptoms at baseline
Correlation between the WPAI : Asthma- Q5 score and the SNOT-22 score | at baseline
  Association between presenteeism and sino-nasal symptoms at baseline
Correlation between the WPAI : Asthma- Q5 score and the AQLQ score | at baseline
  Association between presenteeism and quality of life at baseline
Correlation between the WPAI : Asthma- Q5 score and the daily dose of oral corticosteroids | at baseline
  Association between presenteeism and daily dose of oral corticosteroids at baseline
Correlation between the WPAI : Asthma- Q5 score and the cumulative dose over 6 months of oral corticosteroids | at baseline
  Association between presenteeism and cumulative dose over 6 months of oral corticosteroids at baseline
Correlation between the change in the WPAI : Asthma- Q5 score and in the ACQ-6 score | at baseline and at 6 months
  Association between the change in presenteeism and in asthma control after 6 months of biotherapy
Correlation between the change in the WPAI : Asthma- Q5 score and in the mMRC score | at baseline and at 6 months
  Association between the change in presenteeism and in exercise dyspnea after 6 months of biotherapy
Correlation between the change in the WPAI : Asthma- Q5 score and in FEV1 and R5-R20 | at baseline and at 6 months
  Association between the change in presenteeism and in airways obstruction after 6 months of biotherapy
Correlation between the change in the WPAI : Asthma- Q5 score and in the STAI-Y2 score | at baseline and at 6 months
  Association between the change in presenteeism and in anxiety after 6 months of biotherapy
Correlation between the change in the WPAI : Asthma- Q5 score and in the Nijmegen score | at baseline and at 6 months
  Association between the change in presenteeism and in hyperventilation symptoms after 6 months of biotherapy
Correlation between the change in the WPAI : Asthma- Q5 score and in the SNOT-22 score | at baseline and at 6 months
  Association between the change in presenteeism and in sino-nasal symptoms after 6 months of biotherapy
Correlation between the change in the WPAI : Asthma- Q5 score and in the AQLQ score | at baseline and at 6 months
  Association between the change in presenteeism and in quality of life after 6 months of biotherapy
• Correlation between the change in the WPAI : Asthma- Q5 score and in the daily dose of oral corticosteroids | at baseline and at 6 months
  Association between the change in presenteeism and in the daily dose of oral corticosteroids after 6 months of biotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Chenivesse, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Calmette Chu Lille, Lille, France